CLINICAL TRIAL: NCT00242320
Title: The JADE Study: A 12-week, Double-blind, Randomized Study to Investigate the Effect of 500 mcg Roflumilast Tablets Once Daily Versus Placebo on Pulmonary Function in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Efficacy and Safety of Oral Roflumilast Taken Once Daily in Patients Older Than 40 Years With Chronic Obstructive Pulmonary Disease (BY217/M2-119)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BY217/M2-119
Record Dates: First submitted 2005-10-19; First posted 2005-10-20 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-09

CONDITIONS: COPD
Keywords: COPD; chronic obstructive pulmonary disease; Roflumilast
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator): Roflumilast 500 µg
  Interventions: Drug: Roflumilast
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Roflumilast; Drug: Placebo

INTERVENTIONS:
Drug: Roflumilast — to investigate the effect of 500 µg Roflumilast tablets once daily versus placebo
Drug: Placebo
  Arms: 2

SUMMARY:
The aim of the study is to compare the effect of roflumilast on lung function in patients with COPD. Roflumilast will be administered orally once daily in the morning at one dose level. The study duration consists of a baseline period (4 weeks) and a treatment period (12 weeks). The study will provide further data on safety and tolerability of roflumilast.

ELIGIBILITY:
Main Inclusion Criteria:

* Written informed consent
* Patients with a history of chronic obstructive pulmonary disease (COPD) as defined by the GOLD criteria (2003)
* FEV1/FVC ratio (post bronchodilator) smaller or equal 70%
* FEV1 (post bronchodilator) 30-80% of predicted
* Fixed airway obstruction
* Current smoker or former smoker (smoking cessation at least one year ago) with a smoking history of at least 10 pack years
* Clinically stable COPD within 4 weeks prior to baseline visit
* Availability of a chest x-ray

Main Exclusion Criteria:

* COPD exacerbation indicated by a treatment with systemic glucocorticosteroids
* Lower respiratory tract infection
* Diagnosis of asthma
* Known alpha-1-antitrypsin deficiency
* Need for long term oxygen therapy defined as longer or equal 16 hours/day
* Clinically relevant abnormal laboratory values suggesting an unknown disease and requiring further clinical evaluation (as assessed by the investigator)
* Known infection with HIV, active hepatitis and/or liver insufficiency (according to the Child Pugh score A or worse)
* Diagnosis or history of cancer
* Clinically significant cardiopulmonary abnormalities
* Pregnancy, breast feeding, oocyte donation or oocyte implantation planned during the trial
* Female patients of childbearing potential, not using reliable method of contraception for the entire study duration, post-menopausal > 1 year or who are not using any other method considered sufficiently reliable by the investigator in individual cases
* Participation in another study (use of investigational product) within 30 days preceding the baseline visit or re-entry of patients already enroled in this trial
* Alcohol or drug abuse
* Inability to follow the study procedures due to e.g., language problems, physiological disorders
* Use of not allowed drugs
* Suspected hypersensitivity to the study medication or rescue medication

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 551 (Actual)
Dates: Start 2005-08; Primary Completion 2007-05 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
mean change from randomization to endpoint in lung function (post bronchodilator) | 12 weeks

SECONDARY OUTCOMES:
mean change from randomization to endpoint in pre and post bronchodilator spirometric parameters | 12 weeks
exacerbation rate | 12 weeks
adverse events | 12 weeks
changes in laboratory values | 12 weeks
changes in vital signs | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (21):
- Hong Kong (2):
  - Altana Pharma/Nycomed, Hong Kong
  - Altana Pharma/Nycomed, Shatin, NT, Hong Kong
- Malaysia (4):
  - Altana Pharma/Nycomed, Jalan Rasah, Seremban
  - Altana Pharma/Nycomed, Kota Bharu / Kelantan
  - Altana Pharma/Nycomed, Kota Kinabalu, Sabah
  - Altana Pharma/Nycomed, Kuala Lumpur
- Philippines (2):
  - Altana Pharma/Nycomed, Manila
  - Altana Pharma/Nycomed, Quezon City
- South Korea (10):
  - Altana Pharma/Nycomed, Anvang-Si, Gveonggi-Do
  - Altana Pharma/Nycomed, Gangwon-do
  - Altana Pharma/Nycomed, Gangwon-Do
  - Altana Pharma/Nycomed, Gwangju
  - Altana Pharma/Nycomed, Gyeonggi-do
  - Altana Pharma/Nycomed, Jiniu-Si. Gveongsangnam-Do
  - Altana Pharma/Nycomed, Jungbuk
  - Altana Pharma/Nycomed, Seoul
  - Altana Pharma/Nycomed, Uijongbu-city, Gveonggi-Do
  - Altana Pharma/Nycomed, Ulsan
- Taiwan (3):
  - Altana Pharma/Nycomed, Kaohsiung City
  - Altana Pharma/Nycomed, Taipei
  - Altana Pharma/Nycomed, Tau-Yuan

REFERENCES:
- See also: BY217-M2-119-RDS-2008-07-09.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4480&filename=BY217-M2-119-RDS-2008-07-09.pdf